CLINICAL TRIAL: NCT03493178
Title: Glutathione in Mild Cognitive Impairment
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Rajagopal V Sekhar, Associate Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H42035: Glutathione in MCI
Record Dates: First submitted 2018-02-22; First posted 2018-04-10 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Glycine; Acetylcysteine; Alanine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MCI-active (Active Comparator): 30 Subjects with MCI will receive N-acetylcysteine and glycine for 12-weeks. ll subjects will be studied at baseline prior to supplementation, after completing 12-weeks of supplementation, and 12-weeks after stopping supplementation (i.e. at 24-weeks). Supplements are only provided for first 12-weeks.
  Interventions: Dietary Supplement: Glycine; Dietary Supplement: N-acetylcysteine (NAC)
- MCI-placebo (Placebo Comparator): 30 subjects will received alanine for 12-weeks. All subjects will be studied at baseline prior to supplementation, after completing 12-weeks of supplementation, and 12-weeks after stopping supplementation (i.e. at 24-weeks). Supplements are only provided for first 12-weeks
  Interventions: Dietary Supplement: Alanine

INTERVENTIONS:
Dietary Supplement: Glycine — Dietary Supplement: glycine will be supplemented in the active arm for 12-weeks
  Arms: MCI-active
Dietary Supplement: N-acetylcysteine (NAC) — Dietary Supplement: NAC will be supplemented in the active arm for 12-weeks
  Arms: MCI-active
Dietary Supplement: Alanine — Dietary Supplement: Alanine will be supplemented in the placebo arm for 12-weeks
  Arms: MCI-placebo

SUMMARY:
Elderly humans have an increased risk of dementia which begins as mild defects in memory called mild cognitive impairment. Glutathione (GSH), a key endogenous antioxidant has been linked to cognition. This exploratory study will investigate mechanisms linked to GSH for cognitive impairment (and improvement) by studying humans with mild cognitive impairment who will be evaluated 12-weeks after receiving either N-acetylcysteine and glycine (GSH precursors), or receiving alanine, and a further 12-weeks after stopping these supplements.

DETAILED DESCRIPTION:
Subjects with MCI will be recruited by written informed consent using forms approved by the Baylor IRB. Subjects will stop nonvitamin supplements for 4wks before screening labs (blood count, HbA1c, glucose, lipid profile, liver profile, blood urea nitrogen, Creatinine, thyroid stimulating hormone, free T4), and for the entire 24wks duration of the study. 60 fasted subjects will have the following measures before and after 12wks of supplementation with cysteine (as N-acetylcysteine) plus glycine vs alanine: (1) Cognitive function using ADCS-PACC (Alzheimer's Disease Co-operative Study-Preclinical Alzheimer's Cognitive Composite which includes Free and Cued Selective Reminding Test, Immediate and Delayed paragraph recall score, Digit-Symbol Substitution Test, Mini mental state examination; (2) Red-cell concentrations of GSH, cysteine, glycine, glutamic acid; plasma malondialdehyde, F2/F3-isoprostanes, sICAM, sVCAM, E-selectin; endothelial function; (3) Mitochondrial glucose oxidation by calorimetry. Measures will be repeated for washout effects 12-wks after stopping supplements.

ELIGIBILITY:
Inclusion Criteria at study entry: (1) Diagnosis of Mild Cognitive Impairment Exclusion Criteria at study entry: (1) hospitalization within past 3 months; (2) known diabetes; (3) creatinine greater than or equal to 1.5 mg/dL; (4) hemoglobin concentration less than 11 g/dL; (5) known liver disease, or AST/ALT greater than or equal to 2x ULN; (6) history of stroke, brain tumor, or active heart failure; (7) history of psychiatric disorders; (8) untreated depression.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-19 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognition | Change between 0-weeks and 12-weeks
  Measured using ADCS-PACC

SECONDARY OUTCOMES:
Concentrations of Glutathione | Change between 0-weeks and 12-weeks
  Measured in red cells
Concentrations of TBARS, F2,F3 isoprostanes | Change between 0-weeks and 12-weeks
  Measured in plasma
Endothelial function markers sICAM, sVCAM, E-selectin | Change between 0-weeks and 12-weeks
  Measured in plasma
Endothelial function | Change between 0-weeks and 12-weeks
  Measured using the EndoPAT system
Mitochondrial fuel oxidation in fasted and fed states | Change between 0-weeks and 12-weeks
  Measured using calorimetry
Insulin resistance | Change between 0-weeks and 12-weeks
  Measured as HOMA-IR

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to anyone outside of investigating team